CLINICAL TRIAL: NCT05933057
Title: Randomised, Double-blind, Placebo-controlled, Multicentre Study to Evaluate the Efficacy, Safety and Tolerability of Givinostat in Non-ambulant Patients With Duchenne Muscular Dystrophy
Brief Title: Efficacy, Safety and Tolerability of Givinostat in Non-ambulant Patients With Duchenne Muscular Dystrophy
Acronym: ULYSSES
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Italfarmaco (Industry)
Collaborators: Fortrea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DSC/14/2357/50; 2023-503521-19 (EudraCT Number); U1111-1295-1799 (Other: Universal Trial Number (UTN)); 1008441 (Other: IRAS ID); 277453 (Other: Health Canada)
Record Dates: First submitted 2023-06-16; First posted 2023-07-06 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: Duchenne Muscular Dystrophy; givinostat
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — givinostat; givinostat hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Givinostat (Experimental): Patients will receive concomitant corticosteroid treatment as part of the standard of care.
  Interventions: Drug: Givinostat
- Placebo (Placebo Comparator): Patients will receive concomitant corticosteroid treatment as part of the standard of care.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Givinostat — Givinostat has to be administered twice daily in a fed state according to a flexible dose regimen based on patient weight. Starting dose could be reduced based on predefined safety rules.
  Other Names: ITF2357
  Arms: Givinostat
Drug: Placebo — Placebo, manufactured to mimic givinostat, has to be administered twice daily in a fed state according to a flexible dose regimen based on patient weight. Starting dose could be reduced based on predefined safety rules.
  Arms: Placebo

SUMMARY:
This is a randomised, double-blind, placebo-controlled, multicentre study to evaluate the efficacy, safety, and tolerability of givinostat in non-ambulant male paediatric (aged 9 to <18 years) patients with DMD. 138 patients will be randomised 2:1 to givinostat or placebo and will be treated for 18 months.

* Planned screening duration: approximately 4 weeks (±14 days)
* Planned treatment duration: 18 months (approximately 72 weeks)
* Planned follow-up duration: 4 weeks (±7 days) (for patients not participating in the long-term safety study)
* Total duration of study participation: up to 83 weeks (ie, 20-21 months)

DETAILED DESCRIPTION:
Duchenne muscular dystrophy is a rare, progressive, debilitating and life-threatening condition for which there is a critical need for novel therapies that are effective and well-tolerated in all DMD patients. Steroids are generally recognised as the standard of care in the general DMD population; however, they are not suitable for all patients.

Givinostat, a HDAC inhibitor, was developed for the treatment of DMD based on: (i) the role that increased HDAC activity is thought to exert in contributing to DMD pathogenesis; and (ii) givinostat's ability to counter the pathophysiological and degenerative mechanisms causing muscle insufficiency in boys with DMD.

This study will evaluate the efficacy, safety, and tolerability of givinostat in non-ambulant patients to further corroborate data from the completed phase 3 pivotal study of givinostat in ambulant patients with DMD (ie, Study DSC/14/2357/48, NCT02851797). Primary Objective of the study is to demonstrate the efficacy of givinostat in reducing muscle decline in non-ambulant DMD patients, as measured by Performance of the Upper Limb (PUL) 2.0. Secondary Objectives of the study are to evaluate the safety and tolerability of givinostat in non-ambulant DMD patients, and to further explore the efficacy of givinostat in non-ambulant DMD patients.

A total of 138 patients are planned for enrolment. Patients will be randomised 2:1 to givinostat or placebo and will be treated for 18 months.

The study will be comprised of:

* A screening period, during which eligibility will be confirmed within 4 weeks (±14 days)
* A baseline visit, during which randomisation will be performed
* A double-blind treatment period, during which patients will receive either givinostat or placebo for 18 months (approximately 72 weeks)
* An end of study visit, occurring at Week 72 (±7 days) at the end of the treatment period. At the end of study visit, all the patients (regardless of treatment arm) will be offered enrolment in the long-term safety study DSC/14/2357/51 (NCT03373968) during which they will receive givinostat.
* A follow-up visit, for those patients not consenting to participation in the long-term safety study, that will occur 4 weeks after the end of study visit (ie, Week 76 ±7 days).

ELIGIBILITY:
Inclusion Criteria:

Patients must satisfy all the following criteria:

1. Children and adolescent males aged ≥ 9 to <18 years at screening (patients ≥ 18 years of age at screening will not be enrolled into the study)
2. Are able to give informed assent and/or consent in writing signed by the patient and/or parent/legal guardian (according to local regulations)
3. A genetic diagnosis of DMD
4. Non-ambulant, defined as being wheelchair bound and:

   1. Unable to perform the 10-meter walk/run test (10MWT), or
   2. Unable to complete the 10MWT in 30 seconds or less, without any support or devices
5. Performance of the Upper Limb test (PUL version 2.0) entry item scores 3 to 6
6. If on medication for DMD-associated cardiomyopathy (eg, ACE inhibitor, β-blocker, diuretics), stable for ≥1 month immediately prior to start of study treatment, if any
7. Stable corticosteroids, defined as:

   1. Receiving systemic corticosteroids for a minimum of 6 months immediately prior to start of study treatment
   2. No significant change in dose or dosing regimen (except for adjustments due to body weight change) for a minimum of 6 months immediately prior to start of study treatment
8. Willing to use adequate contraception. Effective contraceptive methods must be used from randomisation visit through 3 months after the last dose of study drug, and include the following:

   1. True abstinence (ie, absence of any sexual intercourse), when in line with the preferred and usual lifestyle of the patient. Periodic abstinence (eg, calendar, ovulation, post-ovulation, and symptothermal methods) and withdrawal are not acceptable methods of contraception
   2. Condom with spermicide and the female partner must use an effective method of contraception, such as an oral, transdermal, injectable or implanted hormonal contraceptive; intrauterine device; bilateral tubal occlusion, or a diaphragm or a barrier method of contraception in conjunction with spermicidal jelly such as for example cervical cap with spermicide jelly.

Exclusion Criteria:

Patients will be excluded from the study if they satisfy any of the following criteria:

1. Exposure to another investigational drug within 3 months prior to start of study treatment.
2. Have exposure to any dystrophin restoration product (eg, Ataluren, Exon skipping) within 6 months prior to the start of study treatment
3. Having received any gene therapy (eg, AAV Micro-dystrophin delivery) prior to start of study treatment
4. Use of any pharmacologic treatment or supplement (other than corticosteroids), that might have had an effect on muscle strength or function within 3 months prior to the start of study treatment (eg, growth hormone); vitamin D, calcium and any other supplements will be allowed
5. Use of testosterone, unless used as a replacement therapy for the treatment of delayed puberty. The testosterone dose and regimen should be stable within 6 months prior to the start of study treatment, and circulating testosterone levels should be within the normal ranges for the patient's age
6. Elbow-flexion contractures >30° in the dominant arm
7. Inability to perform consistent PUL 2.0 measurement within ±2 points without shoulder domain or within ±3 points with shoulder domain during paired testing at screening
8. Forced Vital Capacity % of predicted <40%
9. Requirement for daytime ventilator assistance (Note: Night ventilator assistance and use of bi-level positive airway pressure therapy is allowed)
10. Episode of respiratory failure within the 8 weeks prior to screening
11. Symptomatic cardiomyopathy or heart failure and/or left ventricular ejection fraction <45%
12. Baseline corrected QT interval using Fredericia's formula (QTcF) >450 msec (as the mean of 3 consecutive readings 5 minutes apart) or history of additional risk factors for torsades de pointes (eg, heart failure, hypokalaemia, or family history of long QT syndrome)
13. Major surgical procedure (including scoliosis surgery) planned within 1 year of the start of study treatment
14. Poorly controlled asthma or underlying lung disease such as bronchitis, bronchiectasis, emphysema, recurrent pneumonia that in the opinion of the Investigator might impact respiratory function
15. Platelets, white blood cells, and/or haemoglobin < lower limit of normal (LLN) at screening (Note: for abnormal screening laboratory test results [<LLN], the platelets count, white blood cell, and haemoglobin will be repeated once; if the repeat test result is still <LLN, the patient should be excluded)
16. Fasting triglycerides >300 mg/dL (3.42 mmol/L) at screening (Note: if the value is >300 mg/dL, the triglycerides will be repeated once; if the repeated test result is still >300 mg/dL, the patient should be excluded)
17. Current or history of liver disease or impairment, including but not limited to a baseline elevated total bilirubin (ie, >1.5 × upper limit of normal [ULN]), unless secondary to Gilbert disease or pattern consistent with Gilbert disease
18. Inadequate renal function, as defined by serum Cystatin C result >2 × ULN (Note: if the value is >2 × ULN, the serum Cystatin C will be repeated once; if the repeated test result is still >2 × ULN, the patient should be excluded)
19. Positive test for hepatitis B surface antigen, hepatitis C antibody, or human immunodeficiency virus at screening
20. Hypersensitivity to any component of study medication
21. Sorbitol intolerance or malabsorption, or have the hereditary form of fructose intolerance
22. Diagnosis of other uncontrolled neurological diseases or presence of relevant uncontrolled somatic disorders that are not related to DMD, based on Investigator judgement
23. Psychiatric illness or social situations rendering the potential patient unable to understand and comply with the muscle function tests and/or with the study protocol procedures, based on Investigator judgement
24. Have contraindications to MRI scan (eg, claustrophobia, metal implants, or uncontrolled seizure disorder), based on Investigator's judgement.

Ages: 9 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 138 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Change of Performance of Upper Limb 2.0 (PUL) total score at 18 months of treatment of givinostat compared to placebo group. | Baseline and 18 months
  The PUL examines 3 major "dimensions" of upper extremity function: shoulder, middle, and distal functions. It includes 22 scored items; a score of 42 (12 for shoulder; 17 for mid-level, and 13 for distal) indicates the highest level of independent function and 0 the lowest.

SECONDARY OUTCOMES:
Change from baseline of Peak Expiratory Flow percent predicted (PEF%p) at 18 months of treatment of givinostat compared to placebo group | Baseline and 18 months
Change from baseline of Forced Vital Capacity percent predicted (FVC%p) at 18 months of treatment of givinostat compared to placebo group | Baseline and 18 months
Cumulative loss of PUL total score over 18 months of treatment of givinostat compared to placebo group. | Baseline to 18 months
Type, incidence, and severity of treatment-emergent adverse events | Baseline to 18 months
Proportion of patients experiencing treatment-emergent adverse events | Baseline to 18 months
Change from baseline vital signs and clinical laboratory tests | Baseline and 18 months
Change from baseline electrocardiogram and echocardiogram | Baseline and 18 months
Time to assisted ventilation and rate of respiratory infection including duration, severity of respiratory infection and use of antibiotics, of givinostat compared to placebo group. | Baseline to 18 months

OTHER OUTCOMES:
Change from baseline of Fat Fraction of Deltoid and Biceps brachii using Dixon technique at 18 months of treatment of givinostat compared to placebo group | Baseline and 18 months
Proportion of responders of givinostat compared to placebo group | Baseline to 18 months
  Responders are defined as patients who did not change their baseline PUL entry score at the EOS
Change from baseline of shoulder, elbow and distal level domains of PUL at 18 months of treatment of givinostat compared to placebo group | Baseline and 18 months
Change from baseline in muscle strength (eg, elbow flexion) evaluated by hand held myometry at 18 months of treatment of givinostat compared to placebo group | Baseline and 18 months
Change from baseline in grip strength of dominant hand as measured by Jamar Smart Hand dynamometer at 18 months of treatment of givinostat compared to placebo group | Baseline and 18 months
Change from baseline in physical function as measured by Egen Klassifikation (EK) score at 18 months of treatment of givinostat compared to placebo group | Baseline and 18 months
Change from baseline as measured by Motor Function Measure (MFM) at 18 months of treatment of givinostat compared to placebo group | Baseline and 18 months
Change from baseline of Peak Cough Flow (PCF) at 18 months of treatment of givinostat compared to placebo group | Baseline and 18 months
Age at loss of hand-to-mouth function assessed by PUL | Baseline to 18 months
Age at loss of turn in bed ability assessed by EK | Baseline to 18 months
Change from baseline in DMD Upper Limb Patient-Reported Outcome Measures questionnaire scores at 18 months of treatment of givinostat compared to placebo group | Baseline and 18 months
Change from baseline in quality of life (as measured by Paediatric Quality of Life Inventory 4.0 Generic Core and 3.0 Neuromuscular Module) at 18 months of treatment of givinostat compared to placebo group | Baseline and 18 months
Change from baseline in reports of activities of daily living (as measured by Barthel index) at 18 months of treatment of givinostat compared to placebo group | Baseline and 18 months
Pharmacokinetic/Pharmacodynamic Endpoints | Baseline and 18 months
  PK parameters including, but not limited to, Cmax, T1/2, and AUC, will be assessed using sparse sampling. PD parameters will include PUL, FVC, PEF, MFM, and muscle strength

CONTACTS AND LOCATIONS:
Locations (20):
- Universitaire Ziekenhuizen Leuven, Leuven, Belgium
- Canada (4):
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - The University of Western Ontario - Children's Health Research Institute, London, Ontario
  - University of Ottawa - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - University of Toronto - Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario
- France (3):
  - Centre Hospitalier Régional Universitaire de Lille, Lille
  - Centre hospitalier universitaire - Hôpitaux de Marseille, Marseille
  - Hôpital Armand-Trousseau - I-Motion, Paris
- Germany (2):
  - Charite-Universitaetsmedizin Berlin, Berlin
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
- Italy (5):
  - Associazione La Nostra Famiglia - IRCCS Eugenio Medea - Bosisio Parini, Lecco
  - Fondazione Serena Onlus - Azienda Ospedaliera Niguarda Ca' Granda - NeuroMuscular Omnicentre, Milan
  - Università degli Studi di Padova - Azienda Ospedaliera di Padova, Padua
  - Ospedale Pediatrico Bambino Gesù, Roma
  - Policlinico Universitario Agostino Gemelli - Università Cattolica del Sacro Cuore, Roma
- Netherlands (2):
  - Leids Universitair Medisch Centrum (LUMC), Leiden
  - Radboud Universitair Medisch Centrum (Radboudumc), Nijmegen
- United Kingdom (3):
  - Newcastle upon Tyne Hospitals NHS Foundation Trust - Newcastle University, Newcastle upon Tyne, England
  - Oxford University Hospitals NHS Foundation Trust, Oxford, England
  - NHS Greater Glasgow and Clyde - Royal Hospital for Children, Glasgow, Scotland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bettica P, Petrini S, D'Oria V, D'Amico A, Catteruccia M, Pane M, Sivo S, Magri F, Brajkovic S, Messina S, Vita GL, Gatti B, Moggio M, Puri PL, Rocchetti M, De Nicolao G, Vita G, Comi GP, Bertini E, Mercuri E. Histological effects of givinostat in boys with Duchenne muscular dystrophy. Neuromuscul Disord. 2016 Oct;26(10):643-649. doi: 10.1016/j.nmd.2016.07.002. Epub 2016 Jul 11. PMID 27566866
- [Background] Consalvi S, Mozzetta C, Bettica P, Germani M, Fiorentini F, Del Bene F, Rocchetti M, Leoni F, Monzani V, Mascagni P, Puri PL, Saccone V. Preclinical studies in the mdx mouse model of duchenne muscular dystrophy with the histone deacetylase inhibitor givinostat. Mol Med. 2013 May 20;19(1):79-87. doi: 10.2119/molmed.2013.00011. PMID 23552722
- [Background] Mercuri E, Vilchez JJ, Boespflug-Tanguy O, Zaidman CM, Mah JK, Goemans N, Muller-Felber W, Niks EH, Schara-Schmidt U, Bertini E, Comi GP, Mathews KD, Servais L, Vandenborne K, Johannsen J, Messina S, Spinty S, McAdam L, Selby K, Byrne B, Laverty CG, Carroll K, Zardi G, Cazzaniga S, Coceani N, Bettica P, McDonald CM; EPIDYS Study Group. Safety and efficacy of givinostat in boys with Duchenne muscular dystrophy (EPIDYS): a multicentre, randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Neurol. 2024 Apr;23(4):393-403. doi: 10.1016/S1474-4422(24)00036-X. PMID 38508835
- See also: ULYSSES website — https://ulyssesdmd.study/